CLINICAL TRIAL: NCT03865459
Title: The Effect of Watching Relaxing Video on Pain and Anxiety Levels of Female Patients During Cystoscopy: A Randomized Controlled Trial
Brief Title: The Effect of Watching Relaxing Video During Cystoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, Principal Investigator, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 46418926
Record Dates: First submitted 2019-03-04; First posted 2019-03-06 (Actual); Last update posted 2019-03-12 (Actual); Status verified 2019-03

CONDITIONS: Pain; Anxiety; Urological Nursing; Lower Urinary Tract Symptoms
Keywords: anxiety; cystoscopy; female; nursing; pain; video
MeSH Terms: conditions — Pain; Anxiety Disorders; Lower Urinary Tract Symptoms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video group (Experimental): The video group watched relaxing video with a ceiling mounted television during the whole cystoscopy.
  Interventions: Other: Video group
- Control group (No Intervention): The control group received the standard treatment from a surgical technician who works in the cystoscopy during the whole procedure.The control group didn't watch relaxing video during the procedure.

INTERVENTIONS:
Other: Video group — Patients in the video group started to watch the relaxing video about 5-10 minutes before cystoscopy, and continued to watch video during the whole procedure.
  Arms: Video group

SUMMARY:
The cystoscopy procedure may cause pain and anxiety in patients. Since cystoscopy causes more pain in men, studies on pain and anxiety during cystoscopy are more common in men than women. The aim of this study was to evaluate the effect of watching relaxing video during cystoscopy on the pain and anxiety levels of female patients.

DETAILED DESCRIPTION:
Cystoscopy is a safe procedure with low risk of morbidity commonly used to evaluate lower urinary tract symptoms such as hematuria, voiding disorders, irritant bladder symptoms, anatomical disorders. Patients experience pain and anxiety when cystoscope is inserted into the bladder. The various methods (drug or non-drug) are used for pain and anxiety during the cystoscopy. Although there are a lot of studies on male patients, there are limited studies evaluating pain severity in the female patients during urological procedures. In addition, there wasn't found any randomized controlled study for video use from non-drug methods to distract attention in these patients. Based on the study results in the literature, investigators aimed to evaluate the effect of watching relaxing video on the pain and anxiety levels of female patients during rigid cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* female gender
* rigid cystoscopy for the first time

Exclusion Criteria:

* presence of any contraindication for cystoscopy (such as lidocaine allergy, urinary tract infection, and urethra-related anatomical disorders)
* any analgesic used 24 hours before cystoscopy
* manipulations such as Double-J stent placement or removal, and/or bladder biopsy.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
change on pain intensity as measured by Visual Analog Scale | "5-10 minutes before", "during" and "5 minutes after" cytoscopy.
  The average score change on pain intensity as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure pain intensity. The scale is a measuring tool with length of 0-10 cm (0-100 mm). High scores on the scale indicate that pain intensity is high.

SECONDARY OUTCOMES:
score change on anxiety level as measured by State-Trait Anxiety Inventory | "5-10 minutes before" and "5 minutes after" cytoscopy.
  The average score change on anxiety level as measured by State-Trait Anxiety Inventory. This scale is used to measure anxiety. The scores on the scale ranges from 20 to 80. The high scores on the scale indicate that anxiety is high.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ellerkmann RM, Dunn JS, McBride AW, Kummer LG, Melick CF, Bent AE, Blomquist JL. A comparison of anticipated pain before and pain rating after the procedure in patients who undergo cystourethroscopy. Am J Obstet Gynecol. 2003 Jul;189(1):66-9. doi: 10.1067/mob.2003.377. PMID 12861140
- [Background] Ellerkmann RM, McBride AW, Dunn JS, Bent AE, Blomquist JL, Kummer LG, Melick CF. A comparison of anticipatory and postprocedure pain perception in patients who undergo urodynamic procedures. Am J Obstet Gynecol. 2004 Apr;190(4):1034-8. doi: 10.1016/j.ajog.2003.11.006. PMID 15118637
- [Background] Gezginci E, Iyigun E, Kibar Y, Bedir S. Three Distraction Methods for Pain Reduction During Cystoscopy: A Randomized Controlled Trial Evaluating the Effects on Pain, Anxiety, and Satisfaction. J Endourol. 2018 Nov;32(11):1078-1084. doi: 10.1089/end.2018.0491. PMID 30280915
- [Background] Greenstein A, Greenstein I, Senderovich S, Mabjeesh NJ. Is diagnostic cystoscopy painful? Analysis of 1,320 consecutive procedures. Int Braz J Urol. 2014 Jul-Aug;40(4):533-8. doi: 10.1590/S1677-5538.IBJU.2014.04.13. PMID 25251958
- [Background] Kesari D, Kovisman V, Cytron S, Benjamin J. Effects on pain and anxiety of patients viewing their cystoscopy in addition to a detailed explanation: a controlled study. BJU Int. 2003 Nov;92(7):751-2. doi: 10.1046/j.1464-410x.2003.04477.x. PMID 14616460
- [Background] Raheem OA, Mirheydar HS, Lee HJ, Patel ND, Godebu E, Sakamoto K. Does Listening to Music During Office-Based Flexible Cystoscopy Decrease Anxiety in Patients: A Prospective Randomized Trial. J Endourol. 2015 Jul;29(7):791-6. doi: 10.1089/end.2015.0029. Epub 2015 Apr 13. PMID 25630866
- [Background] Soomro KQ, Nasir AR, Ather MH. Impact of patient's self-viewing of flexible cystoscopy on pain using a visual analog scale in a randomized controlled trial. Urology. 2011 Jan;77(1):21-3. doi: 10.1016/j.urology.2010.08.012. Epub 2010 Oct 25. PMID 20974485
- [Background] Walker MR, Kallingal GJ, Musser JE, Folen R, Stetz MC, Clark JY. Treatment efficacy of virtual reality distraction in the reduction of pain and anxiety during cystoscopy. Mil Med. 2014 Aug;179(8):891-6. doi: 10.7205/MILMED-D-13-00343. PMID 25102532
- [Background] Yeo JK, Cho DY, Oh MM, Park SS, Park MG. Listening to music during cystoscopy decreases anxiety, pain, and dissatisfaction in patients: a pilot randomized controlled trial. J Endourol. 2013 Apr;27(4):459-62. doi: 10.1089/end.2012.0222. Epub 2012 Dec 5. PMID 23009573
- [Background] Zhang ZS, Wang XL, Xu CL, Zhang C, Cao Z, Xu WD, Wei RC, Sun YH. Music reduces panic: an initial study of listening to preferred music improves male patient discomfort and anxiety during flexible cystoscopy. J Endourol. 2014 Jun;28(6):739-44. doi: 10.1089/end.2013.0705. Epub 2014 Mar 31. PMID 24548148